CLINICAL TRIAL: NCT01895777
Title: Open-label, Randomized, Parallel-group, Active-controlled, Multi-centre Non-inferiority Study of Dabigatran Etexilate Versus Standard of Care for Venous Thromboembolism Treatment in Children From Birth to Less Than 18 Years of Age
Brief Title: Open Label Study Comparing Efficacy and Safety of Dabigatran Etexilate to Standard of Care in Paediatric Patients With Venous Thromboembolism (VTE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1160.106; 2013-002114-12 (EudraCT Number)
Record Dates: First submitted 2013-07-04; First posted 2013-07-11 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dabigatran; Standard of Care

ARMS (2):
- dabigatran etexilate (Experimental): Dabigatran etexilate capsules, pellets or liquid formulation given BID in an open label fashion for 3 months
  Interventions: Drug: dabigatran etexilate
- standard of care (Active Comparator): Low molecular weight heparin, vitamin K antagonist or fondaparinux prescribed in an open label fashion for 3 months (these medications will not supplied in this study as IMP)
  Interventions: Drug: standard of care

INTERVENTIONS:
Drug: dabigatran etexilate — Age and weight appropriate capsule dose (combination of 50 mg, 75 mg and 110 mg capsules) or pellets or oral liquid formulation
  Arms: dabigatran etexilate
Drug: standard of care — Low molecular weight heparin, vitamin K antagonist or fondaparinux prescribed in an open label fashion for 3 months (these medications will not supplied in this study as IMP)
  Arms: standard of care

SUMMARY:
The main objectives of this large phase IIb/III paediatric study are to assess the efficacy and safety of dabigatran etexilate relative to standard of care and to document the appropriateness of the proposed dabigatran etexilate dosing algorithm for use in patients from birth to less than 18 years of age.

ELIGIBILITY:
Inclusion criteria:

* Male or female subjects 0 to less than 18 years of age at the time of informed consent / assent
* Documented diagnosis of clinically stable VTE (e.g. DVT, PE, central line thrombosis, sinus vein thrombosis) per investigator judgment, initially treated (minimum of 5 to 7 days, but not longer than 21 days) with parenteral anticoagulation therapy, such as unfractionated heparin (UFH) or a low molecular weight heparin (LMWH).
* Clinical indication for at least 3 month of treatment with anticoagulants for the VTE episode defined under the above inclusion criterion.
* Written informed consent provided by the patient's parent or legal guardian and assent provided by the patient (if applicable) at the time of informed consent form (ICF) signature according to local regulations.

Exclusion criteria:

* Conditions associated with an increased risk of bleeding
* Renal dysfunction (eGFR < 50 mL/min/1.73m^2 using the Schwartz formula) or requirement for dialysis. eGFR retesting during the screening period is allowed (once).
* Active infective endocarditis
* Subjects with a heart valve prosthesis requiring anticoagulation.
* Hepatic disease:

Active liver disease, including known active hepatitis A, B or C or, Persistent alanine aminotransferase (ALT) or aspartate transaminase (AST) or alkaline phosphatase (AP) > 3 × upper limit of normal (ULN) within 3 months of screening

* Pregnant or breast feeding females. Females who have reached menarche and are not using a medically accepted contraceptive method per local guidelines. Acceptable methods of birth control must be used in a correct and consistent manner
* Patients in stratum 3 (0 to < 2 years) with gestational age at birth < 37 weeks or with body weight lower than the 3rd percentile
* Anemia (hemoglobin < 80g/L) or thrombocytopenia (platelet count < 80 x 109/L) at screening. Transfusions during the screening period are allowed, provided that a satisfactory hemoglobin or platelet level is attained prior to visit 2
* Patients who have taken prohibited or restricted medication within one week of the first dose of study medication other than medication for prior VTE treatment and P-glycoprotein inhibitors..
* Patients who have received an investigational drug in the past 30 days prior to screening
* Patients who are allergic/sensitive to any component of the study medication including solvent
* Patients or parents/legal guardians considered unreliable to participate in the trial per investigator judgment or any condition which would present a safety hazard to the patient based on investigator judgment
* Patients or parents/legal guardians who are unwilling or unable to undergo or permit repeat of the baseline imaging tests required to confirm thrombus resolution at study day 84 (or eEOT, whichever comes first) or in whom repeating such imaging tests at these pre-specified time points may not be medically in the patient's best interest. Examples may include unwarranted radiation exposure as a result of a repeat CT scan at day 84 for a patient with an isolated case of pulmonary embolism evaluated at baseline solely by a CT scan. In such cases, the baseline radiological assessment (e.g. CT) may be supplemented with an acceptable non-radiological assessment at baseline (e.g. MRI) which could then be repeated at day 84 hence alleviating any potential unwarranted radiation exposure.
* Further exclusion criteria apply

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 267 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (65):
- United States (9):
  - University of California Davis, Sacramento, California
  - University of Miami, Miami, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Virginia Health System, Charlottesville, Virginia
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
- Hospital General de Niños Pedro de Elizalde, CABA, Argentina
- Austria (2):
  - Medical University of Innsbruck, Innsbruck
  - AKH - Medical University of Vienna, Vienna
- Belgium (3):
  - Brussels - UNIV Saint-Luc, Brussels
  - UNIV UZ Gent, Ghent
  - UZ Leuven, Leuven
- Brazil (4):
  - HMCP - Hospital e Maternidade Celso Pierro - PUC-Campinas, Campinas
  - Faculdade de Ciencias Medicas da UNICAMP, Campinas
  - PenSI - Pesquisa e Ensino em Saude Infantil, São Paulo
  - Instituto de Crianca / Hospital das Clínicas-FMUSP, São Paulo
- Canada (3):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- Czechia (6):
  - University Hospital Brno, Brno
  - General Univ.hosp Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava
  - University Hospital Plzen, Plzen-Lochotin, Plzen-Lochotin
  - University Hospital Motol, Prague
- Rigshospitalet, København, Børneonkologisk Afsnit 5002, Copenhagen, Denmark
- TaUH, Pediatric Early Phase Trial Unit, Tampere, Finland
- HOP de la Cavale Blanche, Brest, France
- Germany (2):
  - Universitätsklinikum Essen AöR, Essen
  - Universitätsklinikum Münster, Münster
- "Aghia Sophia" Children's Hospital, Athens, Greece
- University Debrecen Hospital, Debrecen, Hungary
- Shaare Zedek Medical Center, Jerusalem 91031, Jerusalem, Israel
- Italy (2):
  - Università degli Studi "La Sapienza", Roma
  - Ospedale Infantile Regina Margherita, Torino
- Children Intensive Care Hosp,Anaesthesiology Dept,Vilnius, Vilnius, Lithuania
- Mexico (2):
  - Instituto Nacional de Pediatría, México D.F
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Nuevo León
- Norway (2):
  - Haukeland Universitetssykehus, Bergen
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
- Russia (7):
  - Children Rep.Clin.Hosp of MoH,Cardio Vas.surgery Dept, Kazan, Kazan'
  - Science Res.Instit.CV Diseases,Scientific Res.Dept,Kemerovo, Kemerovo
  - Izmilovskaya Child City ClinHosp,Haematological Dept, Moscow, Moscow
  - Child.CityClin.Hos.na.ZA Bashlyaeva MoscowHealth Dep,Cardiol, Moscow
  - St.Petersburg State Pediatric Univ.Ministry of Healthcare RF, Saint Petersburg
  - Reg Clin.Hosp.#1,Healthcare Tyumen Region,Cardiovas.Surgery, Tyument
  - Childr.CityClin.Hos#9,pediatric&Neonatal Neurol.Ekaterinburg, Yekaterinburg
- Hospital Infantil Universitario Niño Jesus, Madrid, Spain
- Sweden (2):
  - Sahlgrenska US, Göteborg, Gothenburg
  - Karolinska Univ. sjukhuset, Solna
- Universitäts-Kinderspital, Zurich, Switzerland
- Taichung Veterans General Hospital, Taichung, Taiwan
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand
- Turkey (Türkiye) (7):
  - Cukurova Universitesi Tip Fakultesi Cocuk Sagligi, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Istanbul Saglik Bilimleri Uni. Kanuni Sultan Suleyman EAH, Istanbul
  - Ege Universitesi Tip Fakultesi Cocuk Hematolojisi Bilim Dali, Izmir
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi, Konya
- Ukraine (2):
  - Reg.Children Hosp.Dnipropetrovsk, Dnipropetrovsk
  - Reg.Children Hosp,Vinnytsia, Vinnytsia

REFERENCES:
- [Derived] Albisetti M, Tartakovsky I, Halton J, Bomgaars L, Chalmers E, Mitchell LG, Luciani M, Nurmeev I, Gorbatikov K, Miede C, Brueckmann M, Brandao LR; Study Investigators. Dabigatran for Treatment and Secondary Prevention of Venous Thromboembolism in Pediatric Congenital Heart Disease. J Am Heart Assoc. 2024 Feb 20;13(4):e028957. doi: 10.1161/JAHA.122.028957. Epub 2024 Feb 13. PMID 38348778
- [Derived] Brandao LR, Tartakovsky I, Albisetti M, Halton J, Bomgaars L, Chalmers E, Luciani M, Saracco P, Felgenhauer J, Lvova O, Simetzberger M, Sun Z, Mitchell LG. Dabigatran in the treatment and secondary prophylaxis of venous thromboembolism in children with thrombophilia. Blood Adv. 2022 Nov 22;6(22):5908-5923. doi: 10.1182/bloodadvances.2021005681. PMID 36150047
- [Derived] Halton J, Brandao LR, Luciani M, Bomgaars L, Chalmers E, Mitchell LG, Nurmeev I, Sharathkumar A, Svirin P, Gorbatikov K, Tartakovsky I, Simetzberger M, Huang F, Sun Z, Kreuzer J, Gropper S, Reilly P, Brueckmann M, Albisetti M; DIVERSITY Trial Investigators. Dabigatran etexilate for the treatment of acute venous thromboembolism in children (DIVERSITY): a randomised, controlled, open-label, phase 2b/3, non-inferiority trial. Lancet Haematol. 2021 Jan;8(1):e22-e33. doi: 10.1016/S2352-3026(20)30368-9. Epub 2020 Dec 5. PMID 33290737
- [Derived] Albisetti M, Biss B, Bomgaars L, Brandao LR, Brueckmann M, Chalmers E, Gropper S, Harper R, Huang F, Luciani M, Manastirski I, Mitchell LG, Tartakovsky I, Wang B, Halton JML. Design and rationale for the DIVERSITY study: An open-label, randomized study of dabigatran etexilate for pediatric venous thromboembolism. Res Pract Thromb Haemost. 2018 Mar 25;2(2):347-356. doi: 10.1002/rth2.12086. eCollection 2018 Apr. PMID 30046738

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-centre, open-label, randomised, parallel-group, active-controlled, non-inferiority trial of dabigatran etexilate (DE) versus standard of care (SoC) in children from birth to less than 18 years of age.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Dabigatran Etexilate: Oral administration of dabigatran etexilate (DE) twice daily. Patients aged ≥8 years: age- and weight-adjusted DE dosing via capsules using 50 milligram (mg), 75 mg, 110 mg, and 150 mg capsules. Patients aged <8 years or for patients who cannot take capsules even if older than 8 (but <12 years of age): age- and weight-adjusted dosing via DE pellets. Patients aged <12 months: age- and weight-adjusted dosing via DE oral liquid formulation (OLF).
- Standard of Care: Investigators decided on SoC treatment at time of randomisation: either low molecular weight heparin (LMWH) or vitamin K antagonists (VKA) or fondaparinux.
Period: Overall Study
Arm/Group | Dabigatran Etexilate | Standard of Care
Started | 177 | 90
Treated | 176 | 90
Completed | 168 | 85
Not Completed | 9 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Not treated | 1 | 0
Not completed — Other reasons | 3 | 2
Not completed — Non-compliance with the CTP | 2 | 1

BASELINE CHARACTERISTICS:
Population: The randomised set (RS) included all randomised patients in the treatment groups to which they were randomised, regardless whether they took trial medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate | Standard of Care | Total
Number analyzed (Participants) | 177 | 90 | 267
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.1 (6.1) | 11.0 (6.1) | 11.1 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 38 | 134
  Male | 81 | 52 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 169 | 86 | 255
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 163 | 82 | 245
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Composite Primary Endpoint
Description: The primary endpoint was the combined endpoint of the proportions of patients with:
  * Complete thrombus resolution
  * Freedom from recurrent VTE
  * Freedom from mortality related to VTE. The events outlined in the above combined primary endpoint were assessed by radiologists or other such qualified clinicians using an appropriate method such as ultrasound, echocardiography, venography, or CT scan, based on the location of the thrombus and the test used to perform the baseline assessment.
  The primary efficacy endpoint contained 3 components. Each component was evaluated separately, and only if the criteria for all 3 components were satisfied, the primary endpoint was considered achieved.
Time Frame: From the time of randomisation until Week 12, 84 days after randomisation including a visit window of 7 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate | Standard of Care
Number analyzed (Participants) | 177 | 90
Participants
  Complete thrombus resolution | 81 | 38
  Freedom from recurrent VTE | 170 | 83
  Freedom from mortality related to VTE | 177 | 89
  Composite endpoint met | 81 | 38
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Standard of Care; The primary analysis of the primary efficacy endpoint used the randomised set, following the intention-to-treat principle, based on adjudication-confirmed data. Age group was used as stratification factor using a Mantel-Haenszel type weighted average of differences; Test type: Non-Inferiority — Non-inferiority margin of 20%; p = 0.0001, Cochran-Mantel-Haenszel — p-value for non-inferiority is actually <0.0001; Difference in Rates = -0.038, 90% CI 2-sided [-0.141 to 0.066] — Difference in rates (SOC - DE)

2. Secondary Outcome: Freedom From Major Bleeding Events (MBEs)
Description: Freedom from major bleeding events (MBEs), defined as either fatal bleeding, clinically overt bleeding associated with a decrease in haemoglobin of at least 20 g/L in a 24-hour period, bleeding that is retroperitoneal, pulmonary, intracranial or otherwise involves the central nervous system, or bleeding that requires intervention in an operating suite.
Time Frame: From first administration of trial medication until last administration of trial medication +6 days (residual effect period). Up to 97 days.
Population: The treated set (TS) includes all patients who were dispensed trial medication and were documented to have taken at least 1 dose of trial medication
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Dabigatran Etexilate | Standard of Care
Number analyzed (Participants) | 176 | 90
Proportion of participants | 0.977 [0.948 to 0.990] | 0.977 [0.929 to 0.993]
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Standard of Care; Time-to event endpoint using Kaplan-Meier estimates based on adjudication-confirmed data. Due to the low event rate of major bleeding, age group stratification was not considered; Test type: Other; Kaplan-Meier estimate; Kaplan-Meier estimate = 0.000, 90% CI 2-sided [-0.032 to 0.032] — Kaplan-Meier estimate of rate difference

3. Secondary Outcome: Steady State Plasma Concentrations of Total Dabigatran at Visit 3
Description: Descriptive statistics for steady state plasma concentrations of total dabigatran etexilate at visit 3
Time Frame: From the time of randomisation until visit 3
Population: The pharmacokinetic set (PKS) included all patients treated with DE who had at least 1 evaluable PK measurement and had no protocol deviations relevant to the evaluation of PK endpoints. Only scheduled visits were considered
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 139
nanogram per milliliter | 79.8 (68.6) [lower limit 68.6]

4. Secondary Outcome: Steady State Plasma Concentrations After at Least 3 Days Following Any Dabigatran Etexilate Dose Adjustment
Description: Descriptive statistics for steady state plasma concentrations of total dabigatran etexilate after at least 3 days following any dabigatran etexilate dose adjustment
Time Frame: From the time of randomisation until Week 12, 84 days after randomisation including a visit window of 7 days.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 49
nanogram per milliliter | 81.7 (54.7) [lower limit 54.7]

5. Secondary Outcome: Frequency of Dose Adjustment During the Treatment Phase
Description: Frequency of dose adjustments (i.e. number of patients with dose adjustment), temporary and permanent discontinuation from therapy, and number of patients with laboratory monitoring requirements for dose
Time Frame: From first administration of trial medication until last administration of trial medication +6 days (residual effect period).
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate | Standard of Care
Number analyzed (Participants) | 176 | 90
Participants
  With dose adjustment | 63 | 56
  With temporary interruption | 25 | 6
  Laboratory monitoring required | 175 | 82

6. Secondary Outcome: Frequency of Patients Switching the Type of Anti-coagulation Therapy Including Dabigatran Etexilate to Standard of Care Treatment and Switching From One Standard of Care Treatment to Another
Description: Frequency of patients switching the type of anti-coagulation therapy including Dabigatran etexilate (DE) to standard of care (SoC) treatment and switching from one standard of care treatment to another.
  For DE arm, only the switch from DE to SoC was counted, while for the SoC arm, all switches among SoC treatments were counted.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate | Standard of Care
Number analyzed (Participants) | 176 | 90
Participants | 22 | 2

7. Secondary Outcome: Freedom From Thrombus Progression at End of Therapy Compared With Baseline
Description: Freedom from thrombus progression at end of therapy compared with baseline, based on adjudication-confirmed data.
Time Frame: From the time of randomisation until Week 12, 84 days after randomisation including a visit window of 7 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate | Standard of Care
Number analyzed (Participants) | 177 | 90
Participants | 148 | 73

8. Secondary Outcome: All Bleeding Events
Description: The number of participants with bleeding events includes major bleeding events (MBEs), clinically relevant non-major (CRNM) bleeding, minor bleeding events, any bleeding events, and the numbers of the combined endpoint of major and CRNM bleeding events was presented, based on adjudication-confirmed data.
Time Frame: From first administration of trial medication until last adminstration of trial medication +6 days (residual effect period). Up to 97 days.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate | Standard of Care
Number analyzed (Participants) | 176 | 90
Participants
  Any bleeding | 38 | 22
  Major bleeding | 4 | 2
  CRNM bleeding | 2 | 1
  Minor bleeding | 33 | 21
  Major and CRNM bleeding | 6 | 3
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Standard of Care; Any bleeding events was analysed as time-to-event endpoint using a stratified Cox proportional hazard model with treatment as a covariate in the model and age group as the stratification factor. A pooling of age groups was performed as no events were observed in certain age group; Test type: Other; Hazard Ratio (HR) = 1.145, 90% CI 2-sided [0.736 to 1.780]

9. Secondary Outcome: All-cause Mortality
Description: Patients being alive at the end of observational period will be censored for all-cause mortality at the date of patients' last date known to be alive, or the date of data cut-off whichever comes first.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Dabigatran Etexilate | Standard of Care
Number analyzed (Participants) | 176 | 90
Participants | 0 | 1
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Standard of Care; All-cause mortality was analyzed as time-to-event endpoint using a stratified Cox proportional hazard model with treatment as a covariate in the model; Test type: Other; p = 0.9976, Cox proportional hazard model; Hazard Ratio (HR) = 69990000, 90% CI 2-sided [0.000 to 999999999] — Upper Limit of the 90% confidence interval was not assessable

10. Secondary Outcome: All Components of the Primary Efficacy Endpoint
Description: Patients with VTE-related death occurring between randomisation to Day 84 + 7 days were considered as not meeting the endpoint. The presence of recurrent VTE(s) was examined throughout the trial, and only the date of first occurrence was used for analysis. Assessment of index VTE status (best overall response) was scheduled on Day 84 ± 7 days (Visit 8) for patients who were alive without an early consent withdraw. In the case a Patient discontinued trial medication prematurely due to any reason the index VTE assessment took place at the early end of treatment visit.
Time Frame: From the time of randomisation until Week 12, 84 days after randomisation including a visit window of 7 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate | Standard of Care
Number analyzed (Participants) | 177 | 90
Participants
  Complete thrombus resolution by Day 84 | 81 | 38
  Recurrent VTE by Day 84 | 7 | 7
  VTE-related death by Day 84 | 0 | 1

11. Secondary Outcome: Assessment of the Acceptability of an Age-appropriate Formulation at End of Therapy (Capsules)
Description: Acceptability was defined as the overall ability and willingness of the patient to use the medicinal product. Questions regarding acceptability were to be answered by the patient and/or parent/caregiver (as applicable) and by the investigator/site staff.
  Investigator questionnaire capsules: What is your impression about the patient's acceptability of DE intake? The score is 1 (good), 2 (satisfactory), 3 (not satisfactory) and 4 (bad).
  Parents questionnaire capsules: How acceptable was the DE treatment for the child? The score is 1 (good), 2 (satisfactory), 3 (not satisfactory) and 4 (bad).
  Patients questionnaire capsules: Was taking the study capsules easy or difficult? The score is 1 (Very easy), 2 (easy), 3 (neither easy nor difficult), 4 (difficult) and 5 (very difficult).
  Scores refers to the end of treatment.
Time Frame: Assessment at the last study visit at day 84 (+- 7 days), or at day of early termination.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Dabigatran Etexilate: Oral administration of dabigatran etexilate (DE) twice daily. Patients aged ≥8 years: age- and weight-adjusted DE dosing via capsules using 50 milligram (mg), 75 mg, 110 mg, and 150 mg capsules.
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 119
Score
  Investigator questionnaire capsules: number analyzed (Participants) | 111
  Investigator questionnaire capsules | 1.0 (0.2)
  Parents questionnaire capsules: number analyzed (Participants) | 14
  Parents questionnaire capsules | 1.0 (0.0)
  Patient questionnaire capsules: number analyzed (Participants) | 92
  Patient questionnaire capsules | 1.6 (0.9)

12. Secondary Outcome: Assessment of the Acceptability of an Age-appropriate Formulation at End of Therapy (Pellets)
Description: Acceptability was defined as the overall ability and willingness of the patient to use the medicinal product. Questions regarding acceptability were to be answered by the patient and/or parent/caregiver (as applicable) and by the investigator/site staff.
  Investigator questionnaire pellets: What is your impression about the patient's acceptability of DE intake? The score is 1 (good), 2 (satisfactory), 3 (not satisfactory) and 4 (bad).
  Parents questionnaire pellets: Do you think that spitting occurs? The score is 1 (Never), 2 (sometimes) and 3 (often).
  Scores refers to the end of treatment.
Time Frame: Assessment at the last study visit at day 84 (+- 7 days), or at day of early termination.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Dabigatran Etexilate: Oral administration of dabigatran etexilate (DE) twice daily. Patients aged <8 years or for patients who cannot take capsules even if older than 8 (but <12 years of age): age- and weight-adjusted dosing via DE pellets.
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 42
Score
  Investigator questionnaire pellets | 1.2 (0.6)
  Parents questionnaire pellets: number analyzed (Participants) | 33
  Parents questionnaire pellets | 1.2 (0.5)

13. Secondary Outcome: Assessment of the Acceptability of an Age-appropriate Formulation at End of Therapy (Oral Liquid Formulation - OLF)
Description: Acceptability was defined as the overall ability and willingness of the patient to use the medicinal product. Questions regarding acceptability were to be answered by the patient and/or parent/caregiver (as applicable) and by the investigator/site staff.
  Investigator questionnaire flavoured OLF: What is your impression about the patient's acceptability of DE intake? The score is 1 (good), 2 (satisfactory), 3 (not satisfactory) and 4 (bad).
  Investigator questionnaire unflavoured OLF: What is your impression about the patient's acceptability of DE intake? The score is 1 (good), 2 (satisfactory), 3 (not satisfactory) and 4 (bad).
  Parents questionnaire flavoured OLF.: Do you think spitting occurs? The score ranges form 1 (never), 2 ( sometimes) to 3 (often).
  Parents questionnaire unflavoured OLF:Do you think spitting occurs? The score ranges form 1 (never), 2 ( sometimes) to 3 (often).
  Scores refers to the end of treatment.
Time Frame: Assessment at the last study visit at day 84 (+- 7 days), or at day of early termination.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Dabigatran Etexilate: Oral administration of dabigatran etexilate (DE) twice daily. Patients aged <12 months: age- and weight-adjusted dosing via DE oral liquid formulation (OLF).
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 14
Score
  Investigator questionnaire flavoured OLF: number analyzed (Participants) | 7
  Investigator questionnaire flavoured OLF | 1.6 (0.8)
  Investigator questionnaire unflavoured OLF: number analyzed (Participants) | 5
  Investigator questionnaire unflavoured OLF | 1.2 (0.4)
  Parents questionnaire flavoured OLF: number analyzed (Participants) | 7
  Parents questionnaire flavoured OLF | 1.4 (0.5)
  Parents questionnaire unflavoured OLF: number analyzed (Participants) | 5
  Parents questionnaire unflavoured OLF | 1.8 (0.4)

ADVERSE EVENTS:
Time Frame: For DE patients all AEs recorded between first dabigatran etexilate (DE) intake until 6 days after the last administration of dabigatran etexilate. For patients in standard of care arm, all AEs occurred between the first drug intake of standard of care (SOC) until 6 days after the last administration of any standard of care. The Open-label treatment period with DE or SOC is from vist 2 defined as day 0 up to 84 days.
Description: The treated set (TS) includes all patients who were dispensed trial medication and were documented to have taken at least 1 dose of trial medication
Arm/Group | Dabigatran Etexilate | Standard of Care
All-Cause Mortality (participants affected / at risk) | 2/176 | 2/90
Serious Adverse Events (participants affected / at risk) | 25/176 | 18/90
Other Adverse Events (participants affected / at risk) | 59/176 | 16/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dabigatran Etexilate (N=176) | Standard of Care (N=90)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Papilloedema (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (3) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (2) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis haemorrhagic (Gastrointestinal disorders) | 1 (2) | 0 (0)
Implant site necrosis (General disorders) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 1 (1)
Meningitis herpes (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Wound sepsis (Infections and infestations) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 3 (3)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhagic infarction (Vascular disorders) | 0 (0) | 1 (1)
Post thrombotic syndrome (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Takayasu's arteritis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dabigatran Etexilate (N=176) | Standard of Care (N=90)
Diarrhoea (Gastrointestinal disorders) | 9 (11) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 10 (10) | 0 (0)
Vomiting (Gastrointestinal disorders) | 14 (18) | 1 (1)
Pyrexia (General disorders) | 11 (12) | 3 (3)
Nasopharyngitis (Infections and infestations) | 11 (12) | 7 (7)
Headache (Nervous system disorders) | 17 (26) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 6 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT01895777/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT01895777/SAP_001.pdf